CLINICAL TRIAL: NCT00096434
Title: Phase II Trial of Raf Kinase Inhibitor BAY 43-9006 as Single Oral Agent in Patients With Metastatic Breast Cancer Previously Exposed to Anthracycline and/or Taxane
Brief Title: Sorafenib in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01817; NCI-2012-01817 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000393224; NCCTG-N0336; N0336 (Other: North Central Cancer Treatment Group); N0336 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Sorafenib

ARMS (1):
- Arm I (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with metastatic breast cancer. Sorafenib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the tumor response rate in patients with metastatic breast cancer previously treated with an anthracycline- and/or taxane-containing regimen receiving sorafenib.

II. Assess the toxicity profile of this drug in these patients. III. Determine time to disease progression and survival time of patients treated with this drug.

IV. Correlate pre-treatment levels of activated ERK1/2 with tumor response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months until disease progression and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer

  * Clinical evidence of metastatic disease
* Measurable disease
* HER2-positive or -negative disease

  * If HER2 gene amplified or strongly positive for HER2 by immunohistochemistry, patient must have had prior treatment containing trastuzumab (Herceptin®) unless contraindicated
* Previously treated with anthracycline- and/or taxane-containing regimen in the neoadjuvant, adjuvant, or metastatic setting
* Candidate for first- or second-line chemotherapy for metastatic disease
* Core block or tumor slides of the primary or metastatic tumor available
* No known brain metastases
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-1
* At least 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.5 g/dL
* No evidence of bleeding diathesis
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* PT normal
* PTT normal
* INR normal
* Creatinine ≤ 1.5 times ULN
* Calcium normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* No gastrointestinal tract disease that would preclude taking oral medication
* No active peptic ulcer disease
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to sorafenib or other study agents
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other uncontrolled illness
* See Disease Characteristics
* More than 4 weeks since prior immunotherapy
* No concurrent anticancer immunotherapy
* No concurrent bevacizumab
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease
* No concurrent anticancer chemotherapy
* Prior hormonal therapy in the neoadjuvant, adjuvant, or metastatic setting is allowed
* No concurrent anticancer hormonal therapy
* No prior radiotherapy to ≥ 25% of the bone marrow
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery
* No prior surgical procedure that would affect gastrointestinal absorption
* No other concurrent drugs that target vascular endothelial growth factor (VEGF) or VEGF receptors
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
* No concurrent rifampin
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation (i.e., low-dose warfarin) for venous or arterial devices is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed tumor responses, graded according to RECIST criteria | Up to 5 years
  A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. The tumor response rate is defined as the total number of eligible patients who achieved a complete or partial response according to the RECIST criteria divided by the total number of eligible patients enrolled on study. A 90% confidence interval for the true response rate will be constructed using the Duffy-Santner approach.

SECONDARY OUTCOMES:
Time to progression | Time from registration to disease progression, assessed up to 5 years
  Estimated using the Kaplan-Meier method.
Survival time | Time from registration to death, assessed up to 5 years
  Estimated using the Kaplan-Meier method.
Incidence of adverse events, graded according to the NCI-CTC version 3 | Up to 5 years
  The maximum grade for each type of toxicity will be recorded for each patient at each treatment evaluation. The frequency of each type of toxicity will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Perez, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States